CLINICAL TRIAL: NCT04956536
Title: A Retrospective Study of Anterior Tibial Subluxation in the Setting of Anterior Cruciate Ligament Injury and After Anterior Cruciate Ligament Reconstruction
Brief Title: Anterior Tibial Subluxation in the Setting of ACL-injury and After ACL Reconstruction
Status: Enrolling by invitation | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020433
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: anterior tibial subluxation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Demography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Anterior cruciate ligament-injured patients
  Interventions: Other: Demographic data and MRI images were extracted and analyzed

INTERVENTIONS:
Other: Demographic data and MRI images were extracted and analyzed — Demographic data and MRI images were extracted and analyzed. Related factors for anterior tibial subluxation were examined in anterior cruciate ligament-injured patients.

SUMMARY:
To identify the related factors for anterior tibial subluxation (ATS) on anterior cruciate ligament-injured MRI images.

DETAILED DESCRIPTION:
Demographic data and MRI images of anterior cruciate ligament-injured patients were retrospectively analyzed. Anterior tibial subluxation was measured and factors were examined via univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed anterior cruciate ligament injuries
* Available preoperative MRI images at our hospital

Exclusion Criteria:

* Patients were excluded in the case of under 18 years of age
* Bilateral anterior cruciate ligament injuries
* Concomitant posterior cruciate ligament injuries
* Concomitant collateral ligament injuries
* No access to the preoperative MRI scan at our hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACL-injured patients that had suffered from ACL injury and underwent primary ACL reconstruction between January 1, 2013 and December 31, 2015.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Anterior tibial subluxation | Preoperatively
  Anterior tibial subluxation was measured preoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No